CLINICAL TRIAL: NCT03424356
Title: Comparison of Effects of Low Dose Neuromuscular Blocker Added to Propofol Fentanyl Combination During Lma Procedures in Cystoscopy Patients
Brief Title: Effects of Low Dose Neuromuscular Blocker Usage on Laryngeal Mask Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, associate professor, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 2017/15
Record Dates: First submitted 2017-11-15; First posted 2018-02-07 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Anesthesia
Keywords: LMA; Rocuronium bromur; propofol
MeSH Terms: interventions — Rocuronium; Saline Solution; Sodium Chloride; Fentanyl; Narcotics; Propofol; Hypnotics and Sedatives; Cystoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lma with rocuronium bromide (Experimental): In study group, 2-3 mg/kg propofol, 1mcg/kg fentanyl and 0.15 mg/kg rocuronium bromide will be administered during lma insertion in cystoscopy procedure.
  Interventions: Drug: Rocuronium Bromide; Drug: Fentanyl; Drug: Propofol; Procedure: cystoscopy
- lma with saline solution (Active Comparator): In control group, 2-3 mg/kg propofol, 1 mcg/kg fentanyl and saline(no rocuronium) will be administered during lma insertion in cystoscopy procedure.
  Interventions: Drug: Saline Solution; Drug: Fentanyl; Drug: Propofol; Procedure: cystoscopy

INTERVENTIONS:
Drug: Rocuronium Bromide — 0.15 mg/kg rocuronium bromide
  Other Names: nueromusculer blocker
  Arms: lma with rocuronium bromide
Drug: Saline Solution — 1-2 ml saline solution
  Other Names: saline
  Arms: lma with saline solution
Drug: Fentanyl — 1mcg/kg for induction
  Other Names: narcotic analgesic
Drug: Propofol — 2-3mg/kg for anaesthetic induction
  Other Names: hypnotic agent
Procedure: cystoscopy — patients will treated with this surgical procedure
  Other Names: surgical prosedure

SUMMARY:
Cystoscopy is a simple, effective and reliable method in current urological practice. Anesthesia may be required in cystoscopy for therapeutic purpose, however it may not be necessary for diagnostic cystoscopy. General anesthesia, spinal anesthesia, epidural anaesthesia and senile block methods may be performed in therapeutic cystoscopy.

Pain is main reason of failed cystoscopy. Sedo-analgesia and LMA are generally used for diagnostic cystoscopies. LMA is mostly placed under general anesthesia with the combination of propofol-fentanyl and volatile anesthetics. There is no need for muscle relaxant administration in LMA placement, as it is necessary for intubation. However if muscle relaxant is not used, side effects like hiccup, straining, cough, undesirable muscle movement, hypoxia and laryngeal spasm may be observed.

For the improvement of the patient comfort the use of effective muscle relaxants are described in several studies in literature. This study aimed to reveal the quality of anesthesia, hemodynamics, surgical comfort, extra propofol need and recovery time while low dose of muscle relaxant rocuronium was added to propofol-fentanyl combination for LMA placement.

DETAILED DESCRIPTION:
Cystoscopy is a simple, effective and reliable method in current urological practice for the diagnosis and treatment of urethral and bladder pathologies.

Procedure is frequently used for the placement and replacement (removal) of double J stent in patients with ureteral stones .

Cystoscopy may be used for the investigation of hematuria and dysuria and if needed for diagnostic biopsy as well as for therapeutic purpose in patients with bladder and prostate tumor.

Anesthesia may be required in cystoscopy for therapeutic purpose, however it may not be necessary for diagnostic cystoscopy. General anesthesia, spinal anesthesia, epidural anesthesia and senile block methods may be performed in therapeutic systoscopy. Diagnostic cystoscopies may be performed via sedoanalgesia, local anesthetic spray administration, penile block or without any type of anesthesia. Female patients having short urethra are more compatible for local techniques or for the procedures without anesthesia.

Pain is main reason of failed cystoscopy. Sedoanalgesia and LMA are generally used for diagnostic cystoscopies. LMA is mostly placed under general anesthesia with the combination of propofol-fentanyl and volatile anesthetics. There is no need for muscle relaxant administration in LMA placement, as it is necessary for intubation. However if muscle relaxant is not used, side effects like hiccup, straining, cough, undesirable muscle movement, hypoxia and laryngeal spasm may be observed. Placement of LMA may be difficult or sometimes impossible in some patients with limited mouth opening. These patients may experience complications like pain and burning in the mouth, pain in the ear, hoarse voice, swallowing difficulty because of difficult LMA placement in postoperative period.

For the improvement of the patient comfort the use of effective muscle relaxants are described in several studies in literature. This study aimed to reveal the quality of anesthesia, hemodynamics, surgical comfort, extra propofol need and recovery time while low dose of muscle relaxant rocuronium was added to propofol-fentanyl combination for LMA placement.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients
2. ASA I-II patients
3. Cystoscopy patients
4. patients entubated with lariyngeal mask

Exclusion Criteria:

1. Female patients
2. Asa III-IV patients
3. Surgery duration is more than 2 hours
4. Drug abusers
5. Non compromising patients

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2018-12-04 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
questionnaire | up to first 60 minutes
  The quality of LMA placement with or without neuromusculer drug.

SECONDARY OUTCOMES:
questionnaire | up to first 24 hours
  after the surgery soar throat will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: ayşe ülgey, md, Study Chair — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)